CLINICAL TRIAL: NCT03070496
Title: CoHort of Patients to Identify Biological and Imaging markerS of CardiovascUlar Outcomes in ST Elevation Myocardial Infarction
Brief Title: Multicenter Cohort of STEMI Patients
Acronym: HIBISCUS-STEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0570
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
Keywords: Myocardial infarction; bio-collection; Imaging markers; biomarkers; STEMI; clinical outcomes
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- STEMI cohort (Experimental): Patients recruited in the cohort will have 4 additional interventions compared to the usual follow-up :
  * an additional blood sampling at 6 months
  * an additional electrocardiogram (ECG) at 6 months
  * Magnetic Resonance Imaging (MRI)
  * Quality of life questionnaire
  Interventions: Biological: Blood sampling; Procedure: ECG; Device: MRI; Other: Quality of life questionnaire

INTERVENTIONS:
Biological: Blood sampling — Blood sampling will be performed at 6 months after myocardial infarction to analyse diagnostic and prognostic biomarkers
Procedure: ECG — ECG will be performed at 6 months after myocardial infarction
Device: MRI — MRI will be performed at 1month after myocardial infarction to analyse ventricular remodeling and reperfusion.
Other: Quality of life questionnaire — Patients will pass a quality of life questionnaire at 12 months after myocardial infarction

SUMMARY:
Ischemic heart disease is the leading cause of mortality with 7.2 million of death in industrialized countries (WHO data). Myocardial infarction corresponding to acute occlusion of a coronary artery is the most brutal form and the more severe ischemic myocardial disease. Every year in France, about 60,000 Myocardial infarctions hospitalized, 30,000 are diagnosed remotely and 30,000 are revealed by an inaugural sudden death. Although mortality from myocardial decreased by 30% over the past decade, the prognosis is pejorative and difficult to assess precisely. The management of the patient depends on these factors, and justifies an active search on these topics, including the mechanisms of the deleterious ventricular remodeling, myocardial inflammation, reperfusion injury which determines in particular the evolution to heart failure. Cohorts of patients with myocardial infarction are rare but can be very valuable by their clinical, laboratory and imaging well documented. They are the source of new hypotheses for research or interventions as well as the quality of care assessment tool.

The main objective of this project is to identify new markers: biological and imaging, treatment response and prognosis after acute myocardial infarction.

Secondary objectives of the HIBISCUS-STEMI cohort to establish a clinical database, completed by biological samples and by imaging data that can be used in the following areas:

* Descriptive epidemiology of myocardial infarction and myocardial reperfusion
* Pharmacoepidemiology and treatments observatory: safety, efficacy, indication of treatment in real life, costs
* Assessment of the long-term effect of the treatment on the occurrence of heart failure and sudden death
* Quality of life and personal consequences, family, professional and social myocardial infarction
* Research of new diagnostic and prognostic biomarkers
* Research projects (e.g. risk of developing kidney failure or stroke in patients with myocardial infarction compared to the general population).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Diagnosis of STEMI defined by ST segment elevation ≥ 0.2 mV in 2 contiguous leads on a 12-lead ECG.
* Primary Percutaneous coronary intervention (PCI)

Exclusion Criteria:

* Diagnosis of STEMI not confirmed by angiography
* Refusal to participate in the study or to sign the consent
* Impossibility to give information to the subject about the study
* Lack of medical social coverage
* Obvious contraindication to magnetic resonance imaging (claustrophobia, pacemaker, defibrillator, renal insufficiency, known allergy to a contrast agent)
* Deprivation of civil rights
* participating to another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Heart failure stage | Up to 3 years after myocardial infarction
  Heart failure stage will be assessed thanks to the New York Heart Association (NYHA) classification

SECONDARY OUTCOMES:
Infarct size | 1 month after myocardial infarction
  Infarct size will be measured on MRI
Cardiac enzymes rate | H0 (admission in coronary angiography room)
  Cardiac enzymes rate will be analysed in blood samples
Cardiac enzymes rate | H4 (4 hours after reperfusion)
  Cardiac enzymes rate will be analysed in blood samples
Cardiac enzymes rate | H24 (24 hours after reperfusion)
  Cardiac enzymes rate will be analysed in blood samples
Cardiac enzymes rate | H48 (48 hours after reperfusion)
  Cardiac enzymes rate will be analysed in blood samples
Cardiac enzymes rate | 1 month after myocardial infarction
  Cardiac enzymes rate will be analysed in blood samples
Cardiac enzymes rate | 3 months after myocardial infarction
  Cardiac enzymes rate will be analysed in blood samples
Cardiac enzymes rate | 6 months after myocardial infarction
  Cardiac enzymes rate will be analysed in blood samples
Cardiac enzymes rate | 12 month after myocardial infarction
  Cardiac enzymes rate will be analysed in blood samples
EQ-5D score | 12 month after myocardial infarction
  Patients' quality of life will be evaluated thanks to the EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michel OVIZE, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Hôpital Cardiovasculaire Louis Pradel, Bron
  - CHU Strasbourg, Strasbourg
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paccalet A, Crola Da Silva C, Mechtouff L, Amaz C, Varillon Y, de Bourguignon C, Cartier R, Prieur C, Tomasevic D, Genot N, Leboube S, Derimay F, Rioufol G, Bonnefoy-Cudraz E, Mewton N, Ovize M, Bidaux G, Bochaton T. Serum Soluble Tumor Necrosis Factor Receptors 1 and 2 Are Early Prognosis Markers After ST-Segment Elevation Myocardial Infarction. Front Pharmacol. 2021 Sep 1;12:656928. doi: 10.3389/fphar.2021.656928. eCollection 2021. PMID 34539391